CLINICAL TRIAL: NCT05628701
Title: Colectomy Reconstruction for Ulcerative Colitis In Sweden and England: a Multicenter Prospective Comparison Between Ileorectal Anastomosis and Ileal Pouch-Anal Anastomosis After Colectomy in Patients With Ulcerative Colitis.
Brief Title: Colectomy Reconstruction for Ulcerative Colitis, Ileorectal Anastomosis vs Ileal Pouch-Anal Anastomosis in Ulcerative Colitis.
Acronym: CRUISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Karolinska University Hospital (Other); Göteborg University (Other); University College London Hospitals (Other)
Responsible Party: Principal Investigator, Anton Risto, Principal investigator, Linkoeping University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/124-31/2
Record Dates: First submitted 2022-10-28; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases; Ileostomy - Stoma
Keywords: Ulcerative Colitis,; Colectomy; Reconstruction
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Proctocolectomy, Restorative; Ileostomy

STUDY DESIGN:
Intervention Model Description: The CRUISE study is a prospective, non-randomized, non-blinded, multi-center, controlled trial on satisfaction, QoL, function, and complications between IRA and IPAA and permanent stoma among adult UC patients subjected to subtotal colectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IPAA CRUISE (Experimental): Patients eligible for both operations choosing ileal pouch anal anastomosis.
  Interventions: Procedure: Ileal pouch anal anastomosis (IPAA)
- IRA CRUISE (Experimental): Patients eligible for both operations choosing ileorectal anastomosis.
  Interventions: Procedure: Ileorectal anastomosis (IRA)
- IRA Control (Active Comparator): Patients only eligible for ileorectal anastomosis.
  Interventions: Procedure: Ileorectal anastomosis (IRA)
- IPAA Control (Active Comparator): Patients only eligible for ileal pouch anal anastomosis.
  Interventions: Procedure: Ileal pouch anal anastomosis (IPAA)
- Ileostomy Control (Active Comparator): Patients who decline reconstruction.
  Interventions: Procedure: ileostomy

INTERVENTIONS:
Procedure: Ileorectal anastomosis (IRA) — After subtotal colectomy for ulcerative colitis the patients can either keep their end ileostomy or be reconstructed with an anastomosis (connection) between the ileum and the rectal remnant (Ileorectal anastomosis(IRA))
  Arms: IRA CRUISE; IRA Control
Procedure: Ileal pouch anal anastomosis (IPAA) — The rectum is removed and a pouch constructed with the distal part opf the ileum which in subsequently anastomosed (connected) to the anus(Ileal pouch anal anastomosis (IPAA)).
  Arms: IPAA CRUISE; IPAA Control
Procedure: ileostomy — no reconstruction is performed and the patient is left with his/her ileostomy
  Arms: Ileostomy Control

SUMMARY:
Background There are no prospective trials comparing the two main reconstructive options after colectomy for Ulcerative colitis, ileal pouch anal anastomosis and ileorectal anastomosis. An attempt on a randomized controlled trial has been made but after receiving standardized information patients insisted on choosing operation themselves.

Methods Adult Ulcerative colitis patients subjected to colectomy eligible for both ileal pouch anastomosis and ileorectal anastomosis are asked to participate and after receiving standardized information the get to choose reconstructive method. Patients not declining reconstruction or not considered eligible for both methods will be followed as controls. The CRUISE study is a prospective, non-randomized, multi-center, controlled trial on satisfaction, QoL, function, and complications between ileal pouch anal anastomosis and ileorectal anastomosis.

Discussion Reconstruction after colectomy is a morbidity-associated as well as a resource-intensive activity with the sole purpose of enhancing function, Quality of Life and patient satisfaction. The aim of this study is to provide the best possible information on the risks and benefits of each reconstructive treatment.

ELIGIBILITY:
Inclusion criteria:

* Patients with Ulcerative colitis (UC) aged between 18 and 60
* Scheduled for or have previously undergone subtotal colectomy and ileostomy.
* Patients should have sufficient rectal compliance and controllable inflammation in the rectal using topical Mezalasin only.

Exclusion criteria

* Rectal inflammation of Mayo Score >1
* Poor sphincter function, perianal disease
* Uncertainty regarding UC diagnosis P
* Previous colorectal cancer or severe dysplasia
* Primary Sclerosing Colitis diagnosis
* >2 year since subtotal colectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 2months
  yes/no question if the patient is satisfied with his/her choice of operation
Patient satisfaction | 1year
  yes/no question if the patient is satisfied with his/her choice of operation
Patient satisfaction | 5 years
  yes/no question if the patient is satisfied with his/her choice of operation

SECONDARY OUTCOMES:
SF-36(short form-36 item) | 2 months
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability
SF-36(short form-36 item) | 6 months
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability
SF-36(short form-36 item) | 1 year
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability
SF-36(short form-36 item) | 2 years
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability
SF-36(short form-36 item) | 5 years
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability
Female Sexual Function Index-6 (FSFI-6) | 2months
  6 item questionnaire on female sexual function with total score rangeing from 0-34 with lower scores indicating worse sexual functioning.
Female Sexual Function Index-6 (FSFI-6) | 6months
  6 item questionnaire on female sexual function with total score rangeing from 0-34 with lower scores indicating worse sexual functioning.
Female Sexual Function Index-6 (FSFI-6) | 1 year
  6 item questionnaire on female sexual function with total score rangeing from 0-34 with lower scores indicating worse sexual functioning.
Female Sexual Function Index-6 (FSFI-6) | 2 years
  6 item questionnaire on female sexual function with total score rangeing from 0-34 with lower scores indicating worse sexual functioning.
Female Sexual Function Index-6 (FSFI-6) | 5 years
  6 item questionnaire on female sexual function with total score rangeing from 0-34 with lower scores indicating worse sexual functioning.
International Index of Erectile Function-5 (IIEF-5) | 2 months
  5 item questionnaire on erectile (dys)function rangeing from 5 to 25 with lower scores indicating worse erectile functioning.
International Index of Erectile Function-5 (IIEF-5) | 6 months
  5 item questionnaire on erectile (dys)function rangeing from 5 to 25 with lower scores indicating worse erectile functioning.
International Index of Erectile Function-5 (IIEF-5) | 1 year
  5 item questionnaire on erectile (dys)function rangeing from 5 to 25 with lower scores indicating worse erectile functioning.
International Index of Erectile Function-5 (IIEF-5) | 2 years
  5 item questionnaire on erectile (dys)function rangeing from 5 to 25 with lower scores indicating worse erectile functioning.
International Index of Erectile Function-5 (IIEF-5) | 5 years
  5 item questionnaire on erectile (dys)function rangeing from 5 to 25 with lower scores indicating worse erectile functioning.
Shor health scale (SHS) | 2 months
  IDB specific 4 item qualit of life scale rangeing from 0-24 with higher scores indicating worse quality of life.
Shor health scale (SHS) | 6 months
  IDB specific 4 item qualit of life scale rangeing from 0-24 with higher scores indicating worse quality of life.
Shor health scale (SHS) | 1 year
  IDB specific 4 item qualit of life scale rangeing from 0-24 with higher scores indicating worse quality of life.
Shor health scale (SHS) | 2 years
  IDB specific 4 item qualit of life scale rangeing from 0-24 with higher scores indicating worse quality of life.
Shor health scale (SHS) | 5 years
  IDB specific 4 item qualit of life scale rangeing from 0-24 with higher scores indicating worse quality of life.
Öresland Score | 2 months
  Bowel function score rangeing from 0-17 with higher scores indicating worse functioning.
Öresland Score | 6 months
  Bowel function score rangeing from 0-17 with higher scores indicating worse functioning.
Öresland Score | 1 year
  Bowel function score rangeing from 0-17 with higher scores indicating worse functioning.
Öresland Score | 2 years
  Bowel function score rangeing from 0-17 with higher scores indicating worse functioning.
Öresland Score | 5 years
  Bowel function score rangeing from 0-17 with higher scores indicating worse functioning.
failure | 2 months
  Extirpation of reconstruction or permanant stoma deviation
failure | 6 months
  Extirpation of reconstruction or permanant stoma deviation
failure | 1 year
  Extirpation of reconstruction or permanant stoma deviation
failure | 2 years
  Extirpation of reconstruction or permanant stoma deviation
failure | 5 years
  Extirpation of reconstruction or permanant stoma deviation
reoperations | 2 months
  number of reoperations
reoperations | 6 months
  number of reoperations
reoperations | 1 year
  number of reoperations
reoperations | 2 years
  number of reoperations
reoperations | 5 years
  number of reoperations

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nordenvall, Ass. Prof, Study Chair — Karolinska Institutet
Locations (4):
- Sweden (3):
  - Sahlgrenska Univercity Hospital, Gothenburg
  - Linkoeping University hospital, Linköping
  - Karolinska University Hospital, Solna
- St. Mark's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Risto A, Nordenvall C, Deputy M, Hermanson M, Lindforss U, Block M, Faiz O, Myrelid P. Colectomy reconstruction for ulcerative colitis in Sweden and England: a multicenter prospective comparison between ileorectal anastomosis and ileal pouch-anal anastomosis after colectomy in patients with ulcerative colitis. (CRUISE-study). BMC Surg. 2023 Apr 21;23(1):96. doi: 10.1186/s12893-023-01984-x. PMID 37085812